CLINICAL TRIAL: NCT03602690
Title: Dolutegravir, Darunavir/Ritonavir and Optimized NRTI Recycling as a Third-line Antiretroviral Regimen in Cambodia
Brief Title: Evaluation of Third-line cART Regimen in Cambodia (3DICAM)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 12374 3DICAM
Record Dates: First submitted 2018-07-06; First posted 2018-07-27 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: HIV/AIDS
Keywords: Third-line regimen; Dolutegravir; Darunavir; Cambodia
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — dolutegravir; Darunavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dolutegravir + Darunavir/ritonavir + optimized NRTI (Experimental): All patients will receive ART regimen every day including:
  Dolutegravir 50mg once daily Darunavir/ritonavir 600/100 twice daily Optimized NRTI recycling with lamivudine and one other NRTI (zidovudine or tenofovir or abacavir)
  Interventions: Drug: Dolutegravir + Darunavir/ritonavir + optimized NRTI

INTERVENTIONS:
Drug: Dolutegravir + Darunavir/ritonavir + optimized NRTI — Dolutegravir 50mg once daily Darunavir/ritonavir 600/100 twice daily Optimized NRTI recycling with lamivudine and one other NRTI (zidovudine or tenofovir or abacavir)

SUMMARY:
The study aims to evaluate the virological effectiveness of a third-line regimen combining dolutegravir (DTG), ritonavir-boosted darunavir (DRV/r) and optimized NRTI in Cambodian HIV-infected adults, who failed a protease inhibitors (PI)-based second-line regimen despite 3 months of boosted adherence counseling (BAC).

DETAILED DESCRIPTION:
Each patient will be informed of the objectives and the total duration of the study as well as the benefits and risks to participate. After signature of consent form, Genotyping Resistance Test (GRT) and pre-inclusion samples will be done for all patients with HIV RNA > 1000 copies/mL after 3 months of boosted adherence counselling (BAC). After receiving results of the GRT and the pre-inclusion sample, the technical working group (TWG) of HIV national program will decide to switch the patient to third-line regimen or to continue second-line regimen with new BAC.

PI-based second-line regimen will be continue if 1/ GRT shows sensitivity to ATV 2/ GRT shows sensitivity to at least one of the 3 NRTI recommended in Cambodia (AZT, ABC and TDF). In that case, adherence counselling will be boosted according to the new national guidance and the patient will not be enrolled in the study.

In case of intermediate or fully resistance to ATV/r OR sensitivity to ATV but both resistances to AZT, ABC and TDF and after confirmation of eligibility criteria, patient could be enrolled in the study. A third-line regimen will be started including DRV/r 600/100 twice daily + DTG 50 mg once daily + 3TC 300 mg once daily +/- one fully or intermediate sensitive NRTI among TDF, ABC and AZT. The choice of the last NRTI will be discussed and decided by the TWG according to the HBsAg status, to the result of the GRT and to the medical history of the patient.

At 6 months, plasma HIV-1 RNA will be measured:

* HIV1-RNA < 40 copies/mL and no resistance to DRV at inclusion: a switch to DRV/r 800/100mg once daily will be done and adherence counseling provided to confirm the new dosing with the patient
* HIV1-RNA > 40 copies/mL and/or intermediate or fully resistance to DRV at inclusion: the same regimen will be continued and adherence counseling provided

For all patients, a new virological assessment will be done at 9 and 12 months.

DRV and DTG exposure and pharmacokinetic parameters (Cmax, Cmin and AUC) will be estimated for the 20 first enrolled patients, allowing an intra-patient comparison of the 2 dosing regimens of DRV/r for at least 15 patients.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection
* Failing a NNRTI-based first-line regimen
* Failing a PI-based second-line regimen after 3 months of adherence boosting (HIV RNA > 1000 copies/mL)
* HIV strain intermediate or fully resistant to ATV/r OR sensitive to ATV but both resistant to AZT, ABC and TDF
* For women of childbearing age: acceptance to use effective contraceptive methods
* Informed consent obtained with information sheet given and explained before the inclusion visit and the consent form signed by the participant and the parents or legal guardians for adolescents at the latest the day of the inclusion

Exclusion Criteria:

* History of antiretroviral treatment including darunavir and integrase inhibitor
* Active pregnancy < 12 weeks of amenorrhea and desire of pregnancy during the duration of the study
* Opportunistic infection in acute phase at inclusion including tuberculosis treated since less than one month and/or with no stable clinical condition
* Advanced cirrhosis (Child-Pugh score B or C)
* Creatinine clearance < 50 ml/mn
* Any concomitant medical condition that, according to the clinical site investigator would contraindicate participation in the study
* Concurrent participation in any other clinical study without written agreement of the two study teams

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2018-10-04 (Actual); Primary Completion 2022-04-11 (Estimated); Study Completion 2022-04-11 (Estimated)

PRIMARY OUTCOMES:
Virological effectiveness at 6 months | Month 6
  Proportion of patients with plasma HIV-1 RNA < 40 copies/mL by FDA Snapshot analysis

SECONDARY OUTCOMES:
Virological effectiveness at 12 months | Month 12
  Proportion of patients with plasma HIV-1 RNA < 40 copies/mL by FDA Snapshot analysis at 12 months
Incidence of adverse events (safety) | Month 12
  Incidence of grade 3-4 adverse events (ANRS grading table)
Tolerance | Month 12
  Proportion of patients with permanent study treatment discontinuation during the first year
Adherence to treatment strategy | Month 12
  Proportion of patients with adherence > 90%
Plasmatic drug concentrations | Month 1
  Plasmatic dolutegravir concentrations
Plasmatic drug concentrations | Month 1
  Plasmatic darunavir concentrations

CONTACTS AND LOCATIONS:
Locations (1):
- NCHADS, Phnom Penh, Cambodia

IPD SHARING:
Plan to Share IPD: No